CLINICAL TRIAL: NCT06075342
Title: Research of Intracardiac Hemodynamics and Myocardial Strains of Athlete's Heart
Brief Title: Intracardiac Hemodynamics and Myocardial Strain in Athletes and First Responders
Acronym: IHMS
Status: Completed | Type: Observational
Sponsor: Chengdu Sport University (Other)
Collaborators: Institute of Sports Medicine, General Administration of Sport of China (Unknown)
Responsible Party: Principal Investigator, Ping Yang, Principal Investigator, Chengdu Sport University
Other Study IDs: IHMS; 2019YFF0301704 (Other: National Key Research and Development Program (China))
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Structure and Function; Intracardiac Hemodynamic
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- elite athlete: training year > 10 years and weekly training time > 20 hours
  Interventions: Behavioral: exercise
- casual player: training year < 10 years and weekly training time < 20 hours
  Interventions: Behavioral: exercise
- healthy control: healthy participants with irregular exercise habits
  Interventions: Behavioral: exercise
- first responder: first responders with regular exercise training
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — Exercise intervention according to the training program
  Other Names: exercise training

SUMMARY:
The goal of this observational study is to compare the differences of intracardiac hemodynamics and myocardial strain in athletes with different training levels to adapt to long-term high-level training in rest conditions. The main questions aim to answer are: 1. whether an increase in amplitude and duration of intracardiac hemodynamics and myocardial strain compared with healthy controls; 2. Whether significant correlations exist between the hemodynamic indices and training level.

Participants will be asked to filling out the questionnaire, such as the age, training year (the number of years the athlete has participated in any sport), technical hierarchy (promoted by the Competitive Sports Department of the General Administration of Sport of China, weekly training time in the last 6 months, height, weight, body surface area, heart rate, systolic blood pressure, and diastolic blood pressure; and will be asked to perform an examination of transthoracic echocardiography.

Researchers will compare differences of cardiac structure and function, especially the hemodynamics and myocardial strain to see if training level could affect the cardiac function through hemodynamics and myocardial strain.

ELIGIBILITY:
Inclusion Criteria:

* athletes and healthy control subjects without regular exercise habits;
* no specific medical history or chronic illness.

Exclusion Criteria:

* A previous history of arterial hypertension, diabetes mellitus, heart, kidney, hepatic, infectious, psychiatric, malignant, disorders, taking drugs that can influence ECG intervals, and electrolyte imbalance;
* poor echocardiographic image quality and abnormal segmental ventricular wall movement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: athletes with training year > 10 and WTT > 20, athletes with training year < 10 and WTT < 20, healthy controls with irregular exercise habits
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
intracardiac hemodynamics in mmHg/mm using vector flow mapping | through study completion, an average of 1 year
  intraventricular pressure gradient from left ventricular apex to base
myocardial strain in % using two-dimension tissue tracking | through study completion, an average of 1 year
  left ventricular longitudinal strain

SECONDARY OUTCOMES:
wall shear stress in pascal using vector flow mapping | through study completion, an average of 1 year
  segmental wall shear stress of the left ventricle

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Sport University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes